CLINICAL TRIAL: NCT00224159
Title: Does Statin Initiation Undermine Dietary Behavior?
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Other Study IDs: 00710
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: All English Speaking Adults From the Manhattan VA Clinic Who Have Recently Received Their First Prescription for a Statin
Keywords: Statin therapy; Dietary behavior; Attitudes and beliefs; Self efficacy
MeSH Terms: conditions — Behavior | interventions — Pharmaceutical Preparations

INTERVENTIONS:
Behavioral: Drug and Dietary behavior

SUMMARY:
The purpose of this research is to improve our understanding of the effects that taking cholesterol reducing pills have on dietary behavior as well as other health related behaviors

DETAILED DESCRIPTION:
This study explores the impact of initiating statin therapy on subsequent dietary as well as other lifestyle beliefs, attitudes and behaviors.

Specific aims:

1. To test whether the initiation of statin therapy increases dietary saturated fat intake among statin naive patients.
2. To determine what role attitudes, beliefs, expectations, motivation, intention and self-efficacy regarding drug or diet therapy may play in observed changes in dietary behavior after starting statin therapy.

ELIGIBILITY:
Inclusion Criteria:

All English-speaking adults who have recently (within 1 week)received their first prescription for a statin will be eligible.

Exclusion Criteria:

Will include a history of any of the following:

1. Prior CVD (myocardial infarction, angina, angioplasty, stroke, CABG. or arterial bypass surgery)
2. Diabetes patients
3. Psychiatric patients
4. AIDS patients
5. Substance abuse patients
6. Prior cholesterol lowering medication use
7. Inability to complete the interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All English-speaking adults who have recently (within 1 week)received their first prescription for a statin will be eligible.
Sampling Method: Probability Sample
Enrollment: 100
Dates: Start 2005-02; Study Completion 2006-06

PRIMARY OUTCOMES:
How drug or dietary therapy may play a role in dietary behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Natarajan, MD, MSc, Principal Investigator — Weill Medical College of Cornell University; Devin Mann, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The New York Presbyterian Hospital-Weill Medical Center, New York, New York, United States